CLINICAL TRIAL: NCT06406491
Title: Application Observation of Passive Microprocessor-controlled Knees vs. Active Microprocessor-controlled Knees After Transfemoral Amputation
Brief Title: Passive Microprocessor-controlled Knees vs. Active Microprocessor-controlled Knees After Transfemoral Amputation
Status: Recruiting | Type: Observational
Sponsor: Median (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Johannes Schroeter, Clinical Director and Head of Orthopaedic Department, Median
Other Study IDs: Intuy2024
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Amputation
Keywords: transfemoral amputation; prosthetic user; microprocessor-controlled knee; functional outcomes; patient-reported outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Baseline measurements for all subjects is carried out with their own passive microprocessor-controlled knee prosthesis. After 4 weeks of use of active microprocessor-controlled knee, second measurement is carried out. All subjects follow the same study path.
  Interventions: Device: active microprocessor-controlled knee

INTERVENTIONS:
Device: active microprocessor-controlled knee — Active microprocessor-controlled knees are motorized prosthesis, actively supporting the users while walking, getting up, and climbing stairs.

SUMMARY:
This study investigates prosthetic users´ report of passive microprocessor-controlled knees (pMPK) vs. active microprocessor-controlled knees (aMPK). Outcome measurements are assessed at baseline with the pMPK and after 4 weeks of continuous use of aMPK. Measurements consists of functional outcomes, as well as patient-reported outcomes.

DETAILED DESCRIPTION:
The Intuy Knee, an active electronic microprocessor-controlled prosthesis, aims to improve symmetry in joints, torque, and muscle activation compared to passive prostheses. Furthermore, it provides benefits of active prostheses in terms of weight distribution, stair climbing ease, and reduced oxygen consumption. However, there's a lack of research on subjective evaluation by participants. Thus, the study aims to compare the Intuy Knee with passive prostheses regarding functional outcomes and patient-reported outcomes (PROMs).

The target group includes individuals with transfemoral amputation or knee disarticulation, aged 18 and above, with anticipated moderate to high mobility levels, and currently using an electronic prosthetic knee. The study plans to enroll participants nearing the end of their prosthetic cycle, allowing for comparison between different prosthetic options.

Key objectives include comparing walking distance, stair climbing, and hill ascent between passive and active prostheses, as well as evaluating mobility, daily functionality, quality of life, and fear of falling.

The study design is prospective with a pre-post design, aiming for an intra-individual comparison between active and passive prostheses. It outlines inclusion and exclusion criteria, study procedures, and discontinuation criteria for both individual and overall study termination.

ELIGIBILITY:
Inclusion Criteria:

* transfemoral amputation or knee-disarticulation
* passive microprocessor-controlled knee
* resupply with new prosthesis within the next few months
* K-Level 2 or 3
* body weight no more than 125 kg
* German speakers

Exclusion Criteria:

* age less than 18 years
* unable to give informed consent
* body weight more than 125 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with transfemoral amputation or knee-disarticulation. The subjects are already provided with a passive microprocessor-controlled knee, but are about to receive their final prosthesis (6 months past interim prosthesis) or they are entitled for a new prosthesis (usually after 5 years with the same prosthesis). Subjects have a moderate (K2-K3) mobility grade.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | baseline (t1), after 4 weeks (t2)
  Subject walks for 6 minutes a defined track and covered track is reported as meters
Stair Assessment Index (SAI) | baseline (t1), after 4 weeks (t2)
  Subjects walks up and down a stair 3 times, the investigator rates the performance on a scale from 0 (cannot to/refused to do) - 13 (without rail or assisstive device, step-over-step pattern) points
Hill Assessment Index (SAI) | baseline (t1), after 4 weeks (t2)
  Subjects walks up and down a hill 3 times, the investigator rates the performance on a scale from 0 (cannot to/refused to do) - 11 (even step without assisstive device) points

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | baseline (t1), after 4 weeks (t2)
  Subjects gets up from a chair, walks 3 metres, turns, walks back to the chair, and sits down. The investigator records the time (seconds).
Amputee Mobility Predictor with Prosthesis (AMP-PRO) | baseline (t1), after 4 weeks (t2)
  Functional Assessment of 21 different tasks and evaluations. The investigator rates each tasks and sums up the score (min. 0; max. 47 points)
Prosthetic Limb User´s Survey of Mobility (PLUS-M) | baseline (t1), after 4 weeks (t2)
  Questionnaire assessing users´mobility with 12 questions. Users rate their answers from 0 ("not able to") to 5 (without any difficulties") points. Results are presented as t-scores from 23.1 - 65.7
EuroQol (EQ5D-5L) questionnaire | baseline (t1), after 4 weeks (t2)
  Questionnaire assessing users´ quality of life. Users rate 5 statements with 1 ("no agreement") to 5 ("complete agreement") points. In addition, the users rate their perceived health on a scale from 0% - 100%. Results are presented as health utility scores. Minimum score is -0.661, maximum score is 1.
Locomotor Capability Index 5 (LCI 5) | baseline (t1), after 4 weeks (t2)
  Questionnaire assessing users´ locomotor abilities. Users rate statements with 0 ("no") to 4 ("yes, without any further assistance) points. Results are presented as "basic activities" (7questions) and "advanced activities" (7 questions). Minimum score is 0 points, maximum score is 28 points for each of the two categories.
Fear of falling | baseline (t1), after 4 weeks (t2)
  Subjects rate their fear of falling indoors and outdoors on a visual analogue scale. Minimum score is 0 (no fear) and maximum score is 10 (maximum fear).

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Schröter, Dr. med., Principal Investigator — MEDIAN Reha-Center Wiesbaden Sonnenberg
Locations (1):
- MEDIAN Clinics, Wiesbaden, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Probsting E, Blumentritt S, Kannenberg A. [Changes in the Locomotor System as a Consequence of Amputation of a Lower Limb]. Z Orthop Unfall. 2017 Feb;155(1):77-91. doi: 10.1055/s-0042-112821. Epub 2016 Sep 15. German. PMID 27632668
- [Background] Hunt GR, Hood S, Gabert L, Lenzi T. Can a powered knee-ankle prosthesis improve weight-bearing symmetry during stand-to-sit transitions in individuals with above-knee amputations? J Neuroeng Rehabil. 2023 May 2;20(1):58. doi: 10.1186/s12984-023-01177-w. PMID 37131231
- [Background] Hunt GR, Hood S, Gabert L, Lenzi T. Effect of Increasing Assistance From a Powered Prosthesis on Weight-Bearing Symmetry, Effort, and Speed During Stand-Up in Individuals With Above-Knee Amputation. IEEE Trans Neural Syst Rehabil Eng. 2023;31:11-21. doi: 10.1109/TNSRE.2022.3214806. Epub 2023 Jan 30. PMID 36240032
- [Background] Ledoux ED, Goldfarb M. Control and Evaluation of a Powered Transfemoral Prosthesis for Stair Ascent. IEEE Trans Neural Syst Rehabil Eng. 2017 Jul;25(7):917-924. doi: 10.1109/TNSRE.2017.2656467. Epub 2017 Jan 20. PMID 28113346